CLINICAL TRIAL: NCT07323095
Title: A Phase 2, International, Multicenter, Randomized, Double-blind, Parallel-group Trial to Evaluate the Efficacy and Safety of ABP-671 in Subjects With Chronic Kidney Disease and Hyperuricaemia
Brief Title: Evaluate the Efficacy and Safety of ABP-671 in Subjects With Chronic Kidney Disease and Hyperuricaemia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Atom Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABP-671-202
Record Dates: First submitted 2025-12-08; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ABP-671 plus febuxostat Group 1 (Active Comparator): Investigators may consider the use of urine alkalinizing agents on an as-needed basis according to the subject's specific condition and standard clinical practice
  Interventions: Drug: ABP-671 plus febuxostat Group 1
- ABP-671 plus febuxostat Group 2 (Active Comparator): Investigators may consider the use of urine alkalinizing agents on an as-needed basis according to the subject's specific condition and standard clinical practice
  Interventions: Drug: ABP-671 plus febuxostat Group 2
- ABP-671 Group (Experimental): Investigators may consider the use of urine alkalinizing agents on an as-needed basis according to the subject's specific condition and standard clinical practice
  Interventions: Drug: ABP-671 Group

INTERVENTIONS:
Drug: ABP-671 plus febuxostat Group 1 — ABP-671 Dose 1 + Febuxostat Dose 1-tablets(PO)
  Arms: ABP-671 plus febuxostat Group 1
Drug: ABP-671 plus febuxostat Group 2 — ABP-671 Dose 2 + Febuxostat Dose 2-tablets(PO)
  Arms: ABP-671 plus febuxostat Group 2
Drug: ABP-671 Group — ABP-671 Dose 2 + Febuxostat placebo-tablets(PO)
  Arms: ABP-671 Group

SUMMARY:
This is a phase 2, international, multicenter, randomized, double blind, parallel group trial to evaluate the efficacy and safety of ABP-671 in subjects with CKD and hyperuricaemia, to preliminarily evaluate the efficacy of ABP-671 in the treatment of subjects with CKD and hyperuricemia, primary Efficacy Endpoint is change in UACR from baseline to Week 28

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-75 years , who voluntarily participate in this clinical trial, understand and comply with the procedures stipulated in this study
* Patients who have been diagnosed with CKD based on Clinical Practice Guideline
* During screening, body mass index (BMI) was ≥18.0 and ≤ 40.0 kg/m2
* The sUA levels > 420 μmol/L (7.0 mg/dL)

Exclusion Criteria:

* History of renal transplantation
* The 24-hour urinary protein ≥ 3.5 g/day
* Liver function abnormality: aspartate aminotransferase or alanine aminotransferase, or alkaline phosphatase > 3 times the upper limit of normal value (ULN)
* Subjects with mental disorders who are unable to communicate normally with the investigator
* Subjects who have participated in another clinical study during the screening period are within 30 days of the last dose of the study drug in another study
* The investigator judged that the subject was not suitable for participation in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
The change in the urine albumin-to-creatinine ratio (mg/g) as reported in the laboratory report compared to the baseline | Week 28

SECONDARY OUTCOMES:
The change in the urine albumin-to-creatinine ratio (mg/g) as reported in the laboratory report compared to the baseline | Week 16
Incidence of treatment-emergent adverse events (Safety and Tolerability) | Week 28
  Incidence of treatment-emergent adverse events (TEAEs), including AEs of special interest (AESIs), serious AEs (SAEs), and AEs leading to study treatment discontinuation

CONTACTS AND LOCATIONS:
Locations (8):
- Genesis Research services, Newcastle, New South Wales, Australia
- China (7):
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital , affiliated with the Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang